CLINICAL TRIAL: NCT06113822
Title: Investigation of The Effect of Body Mass Index and Anxiety on Masseter Muscle Thickness on Ultrasonography
Status: Completed | Type: Observational
Sponsor: Oguzhan Deveci (Other)
Responsible Party: Sponsor-Investigator, Oguzhan Deveci, Principal Investigator, DDS, Firat University
Organization: Firat University (Other)
Other Study IDs: FiratCerrahi
Record Dates: First submitted 2023-10-30; First posted 2023-11-02 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Anxiety
Keywords: anxiety; body mass index; masseter muscle; obesity; ultrasonography
MeSH Terms: conditions — Anxiety Disorders; Obesity | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control Group: Without Anxiety - Normal BMI 15 patient nonanxiety group (HAD scores ranging from 0 to 10) body mass index is normal between 18.5-24.9
  Interventions: Device: ultrasonography
- 1st working group: High BMI & Anxiety Normal 19 Patient nonanxiety group (HAD scores ranging from 0 to 10) Those with a high body mass index are between 25 and 29.9.
  Interventions: Device: ultrasonography
- 2st working group: Normal BMI & High Anxiety (15 patients) having anxiety group (HAD scores ranging from 11 to 21) body mass index is normal between 18.5-24.9
  Interventions: Device: ultrasonography
- 3st working group: High BMI & High Anxiety (19 patients) having anxiety group (HAD scores ranging from 11 to 21) Those with a high body mass index are between 25 and 29.9.
  Interventions: Device: ultrasonography

INTERVENTIONS:
Device: ultrasonography — We used ultrasonography to measure the patients' masseter muscle thickness. Measurements were performed simultaneously for both the right and left sides using a high frequency linear scanning probe (13-6 MHz) of an ultrasound device (Fujifilm Sonosite Edge II). In order to prevent possible artifacts and oblique imaging, the probe was kept perpendicular to the skin surface, and the distance between the location of the hyperechoic linear appearance of the mandibular and temporal bone in the transverse section and the muscular fascia were measured.

SUMMARY:
The aim of this study is to determine the effect of body mass index (BMI) and anxiety on masseter muscle thickness by using ultrasonography.

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of body mass index (BMI) and anxiety on masseter muscle thickness by using ultrasonography.

A total of 68 patients were included in this study. Height and weight of the patients were measured. BMI was calculated. The Control Group Without Anxiety - Normal BMI (15 patients) was composed of patients in general. Working groups were formed as High BMI & Anxiety Normal (19 patients), Normal BMI & High Anxiety (15 patients), and High BMI & High Anxiety (19 patients). The Hospital Anxiety Depression Scale (HADS) was applied to the participants. Muscle thickness measurements were first measured by using the high-frequency linear scanning probe of an ultrasound device to measure the contraction and relaxation of the right masseter muscle. Then, the contraction and relaxation of the left masseter muscle was measured.

ELIGIBILITY:
Inclusion Criteria:

* The study group consisted of individuals between the ages of 18 and 45 who, according to an examination of the masseter muscles under the 'Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD),' had the presence of pain in at least one region in the palpation made from three regions (origin, center, attachment zone) or had pain in chewing muscles in the preceding month.

Exclusion Criteria:

* Exluded from the study where those who had experienced any systemic discomfort from the study group, those who had undergone acute temporomandibular joint trauma, those who had experienced early occlusion of the teeth, those who were using any moving dental prosthesis, those with clenching habits, those who use cigarette-alcohol, those with temporomandibular joint discomfort, and those with unilateral chewing habits.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals in the Turkish population aged 18-45
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
BMI and anxiety | 2022
  Increased BMI and the presence of anxiety cause thickening of the masseter muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- Firat University, Elâzığ, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I'm undecided